CLINICAL TRIAL: NCT07143799
Title: Scalp Block Versus General Anesthesia in Patients Undergoing Evacuation of Subdural Hematoma Via Burr Hole
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Housny Elsayed, Resident , Anesthesia , Surgical Icu , Pain management Faculty of Medicine Sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-8-8MS
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural | interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Group A will receive general anesthesia (Active Comparator): Induction of general anesthesia will be done by IV propofol 2-2.5 mg / kg and IV fentanyl lug/kg. After IV Cis-atracurium 0.15mg/kg, endotracheal intubation will be done.
  Interventions: Drug: Cisatracurium
- Group B patients will receive scalp block (Active Comparator): The scalp block will target six pairs of sensory nerves that innervate the scalp: the supraorbital nerve, supratrochlear nerve, auriculotemporal nerve, zygomaticotemporal nerve, greater occipital nerve, and lesser occipital nerve.Local anesthetic (2% lidocaine and bupivacaine) will be infiltrated at specific anatomical landmarks corresponding to the course of each nerve
  Interventions: Other: scalp block

INTERVENTIONS:
Drug: Cisatracurium — Induction of general anesthesia will be done by IV propofol 2-2.5 mg / kg and IV fentanyl lug/kg. After IV Cis-atracurium 0.15mg/kg, endotracheal intubation will be done.
  Arms: 'Group A will receive general anesthesia
Other: scalp block — The scalp block will target six pairs of sensory nerves that innervate the scalp: the supraorbital nerve, supratrochlear nerve, auriculotemporal nerve, zygomaticotemporal nerve, greater occipital nerve, and lesser occipital nerve. Local anesthetic (2% lidocaine and bupivacaine) will be infiltrated at specific anatomical landmarks corresponding to the course of each nerve.
  Arms: Group B patients will receive scalp block

SUMMARY:
this study amis to compare between Scalp block versus general anesthesia in patients undergoing evacuation of subdural hematoma via burr hole.

ELIGIBILITY:
Inclusion Criteria

* Age from 18 to 75 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status II-III.
* Patients with subdural hematoma undergoing burr-hole evacuation

Exclusion Criteria:

* Patients with a history of known sensitivity to study drugs.
* Glasgow Coma Scale (GCS) <8
* Impaired coagulation profile.
* Any degree of heart block.
* Infection at site of injection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
The aim of this prospective randomized study is to compare Scalp block versus general anesthesia in patients undergoing evacuation of subdural hematoma via burr hole. | 24 hours after operation
  Post operative scale by The Glasgow Coma Scale (GCS) and post operative hemodynamics.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Scruton TJ. Updates on the diagnosis and management of subdural hematoma. JAAPA. 2024 Aug 1;37(8):9-15. doi: 10.1097/01.JAA.0000000000000055. Epub 2024 Jul 25. PMID 38980290
- [Background] Knopman J, Link TW, Navi BB, Murthy SB, Merkler AE, Kamel H. Rates of Repeated Operation for Isolated Subdural Hematoma Among Older Adults. JAMA Netw Open. 2018 Oct 5;1(6):e183737. doi: 10.1001/jamanetworkopen.2018.3737. PMID 30646255
- [Background] Sharma R, Rocha E, Pasi M, Lee H, Patel A, Singhal AB. Subdural Hematoma: Predictors of Outcome and a Score to Guide Surgical Decision-Making. J Stroke Cerebrovasc Dis. 2020 Nov;29(11):105180. doi: 10.1016/j.jstrokecerebrovasdis.2020.105180. Epub 2020 Aug 7. PMID 33066943